CLINICAL TRIAL: NCT03026374
Title: Effect of a Mentor-based, Supportive-expressive Program on Survival in Metastatic Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zeng Jie Ye, Doctor, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZYZC20160901; ZYZC20160901 (Other Grant/Funding Number: State Administration of Traditional Chinese Medicine)
Record Dates: First submitted 2017-01-14; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Breastcancer
Keywords: psychosocial support; resilience; metastatic breast cancer; survival; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): The BRBC program consists of education and group discussion, and lasted for 12 months. Women in IG attended weekly meetings lasting for 120 minutes. Education took approximately 45 minute. Qualified professionals from various disciplines were invited to provide lessons to ensure the quality of the educational sessions. The group discussion followed the presentation and began with mentors sharing their experience with the topic, followed by participant discussions regarding life changes since diagnosis (e.g., physical, emotional, social, spiritual). Each group consisted of 7-9 patients and 3 leaders (2 mentors and 1 facilitator, including a clinical psychologist, nurse clinician, or social worker). The time of group discussion varied from 45-75 minutes. This was intended to foster support among group members,both in and out of sessions.
  Interventions: Behavioral: Be Resilient to Breast Cancer
- control group (No Intervention): patients from both groups were provided medical, social, or psychological care if necessary, as assessed by primary oncologists. Additionally, all patients received an educational brochure about breast cancer every 1 to 2 months, and relaxation therapy was provided to both groups to prevent demoralization from random assignment.

INTERVENTIONS:
Behavioral: Be Resilient to Breast Cancer — This is a supportive-expressive group therapy.
  Other Names: BRBC
  Arms: intervention group

SUMMARY:
Breast cancer is the most prevalent cancer in women and annually accounts for 10% of new malignancies worldwide. In mainland China, approximately 169,000 females are diagnosed with breast cancer every year and constitute 12.25% of the breast cancer incidents worldwide. Additionally, 30% of early breast cancer turns metastatic, which is often incurable. Different from women with early breast cancer, women with metastatic breast cancer(MBC)must receive lifelong treatment, experience higher levels of emotional/physical distress, and feel frequent uncertainty about their health/possible death. They are also challenged to manage distressing adverse effects induced by different adjuvant treatments and experience heavy self-care demands during the transition period from being a patient to being a survivor. Thus, specific interventions to help women with metastatic breast cancer to recover from this traumatic event have been designed, and one of these is supportive-expressive group therapy(SEGT).SEGT has been found to achieve improvement in anxiety, depression, quality of life (QoL), family functioning, and satisfaction with treatment. However, the effect of SEGT on survival is inconsistent. Initial studies examining SEGT have reported a mean survival advantage of 18 months, however, these findings could not later be replicated.Yet, no study has reported a survival disadvantage for those given SEGT. In addition, we found no published articles on the application of SEGT among women with MBC in China. Owing to this dearth of previous research, it is unclear whether this therapy would exhibit positive effects within Chinese culture. Thus, we developed a "Be Resilient to Breast Cancer"(BRBC) program that is culturally tailored for Chinese females with MBC. This program was adapted from SEGT and is designed to increase resilience(defined as the capacity to bounce back after encountering a traumatic event) and QoL, decrease emotional and physical distress(allostatic load), and eventually prolong longevity. To better adapt to Chinese culture, we added education hosted by professional staff (e.g., clinical psychologists, dietician, Chinese medicine practitioner, etc.)in an effort to foster self-efficacy to combat symptoms (such as pain, fatigue, intrusive thoughts, etc.) through knowledge and technics (such as breath control, meditation, etc.),and to help patients gain a sense of control in their life. Second, trained mentors, who were breast cancer survivors themselves, were added to the group discussion to create non-hierarchical, reciprocal relationships through the sharing of experiences with those facing similar challenges. These mentors also provided women with first-hand information about treatment and offered suggestions to combat barriers to recovery.

ELIGIBILITY:
Inclusion Criteria:

* (1) women with confirmed breast cancer, stratified by stage(II,III, and IV),(2) metastases outside of the breast and ipsilateral axilla, and (3) fluent in oral Mandarin or Cantonese.

Exclusion Criteria:

* (1) central nervous system metastases, (2) a history of repeated suicidal behavior, (3) active psychosis or severe character disorder, (4) a life expectancy of less than 3 months(as assessed by primary oncologist), and/or (5)declined to participate in the program

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2017-06; Primary Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
3- and 5-year survival | 3 and 5 years since intervention

SECONDARY OUTCOMES:
allostatic load index(ALI) | baseline, 2 months, 6 months, and 12 months since intervention
  ALI was a composite index measured by 14 indicators from different physiological systems, including body mass index (BMI), waist-hip ratio (WHR), resting pulse(RP), the standard deviation of R-R intervals (SDRR, heartbeat to heartbeat), resting systolicand diastolic blood pressure(SBP and DBP, respectively), white blood cell count (WBC), red blood cell count (RBC), hemoglobin, serotonin, hormone cortisol(HC), C-reactive protein(CRP), interleukin-6 (IL-6) and Cluster of Differentiation 4/ Cluster of Differentiation 8(CD4+/CD8+). These indicators were selected to evaluate the functions of sympathetic nervous system (SNS), parasympathetic nervous system (PNS), hypothalamic pituitary adrenal (HPA), cardiovascular, inflammation, and immunization. If a physical indicator was diagnosed as abnormal (i.e., RP of 107; normal range 60-100), patient would receive 1 point. Higher point totals indicated higher allostatic load. ALI range was from 0(extremely low) to 14(extremely high).
Resilience | baseline, 2 months, 6 months, and 12 months since intervention
  Resilience was measured by the 10 item Conner-Davison Resilience Scale (CD-RISC-10), which is a self-administered questionnaire based on a 5-point scale, with higher scores reflecting more resilience.
Quality of Life | baseline, 2 months, 6 months, and 12 months since intervention
  QoL was measured by QLQ-C30 core questionnaire of the European Organization for Research and Treatment of Cancer (EORTC), which contains 30 items pertaining to different patient QoL aspects.
Anxiety | baseline, 2 months, 6 months, and 12 months since intervention
  Anxiety was measured by the Chinese version of Hospital Anxiety and Depression Scale (HADS), which contains 7 items for anxiety and 7 items for depression, respectively, scored on a 5-point scale. Higher scores indicate higher levels of anxiety.
Depression | baseline, 2 months, 6 months, and 12 months since intervention
  Depression was measured by the Chinese version of Hospital Anxiety and Depression Scale (HADS), which contains 7 items for anxiety and 7 items for depression, respectively, scored on a 5-point scale. Higher scores indicate higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeng Jie Ye, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang MZ, Chen P, Tang Y, Liang YY, Li SH, Hu GY, Sun Z, Yu YL, Molassiotis A, Knobf MT, Ye ZJ. Associations Between Brain Structural Connectivity and 1-Year Demoralization in Breast Cancer: A Longitudinal Diffusion Tensor Imaging Study. Depress Anxiety. 2024 Sep 26;2024:5595912. doi: 10.1155/2024/5595912. eCollection 2024. PMID 40226738
- [Derived] Liang MZ, Zhou J, Chen P, Song YL, Li SH, Liang YY, Hu GY, Hu Q, Sun Z, Yu YL, Molassiotis A, Knobf MT, Ye ZJ. A Longitudinal Correlational Study of Psychological Resilience, Depression Disorder, and Brain Functional-Structural Hybrid Connectome in Breast Cancer. Depress Anxiety. 2024 Nov 18;2024:9294268. doi: 10.1155/2024/9294268. eCollection 2024. PMID 40226657